CLINICAL TRIAL: NCT07359820
Title: A Phase 2, Open-Label, Single-Arm Study of Lirafugratinib in Patients With Previously Treated, Unresectable, Locally Advanced or Metastatic Solid Tumors (Excluding Cholangiocarcinoma) With FGFR2 Fusion or Rearrangement
Brief Title: A Study of Lirafugratinib in Non-CCA Solid Tumors With FGFR2 Fusion or Rearrangement
Acronym: ReFocus202
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELE-4008-202
Record Dates: First submitted 2026-01-16; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: FGFR2 Gene Fusion/Rearrangement; Other Solid Tumors, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lirafugratinib (Experimental): Treatment with standard dose of lirafugratinib
  Interventions: Drug: Lirafugratinib

INTERVENTIONS:
Drug: Lirafugratinib — Lirafugratinib is an oral inhibitor of FGFR2
  Other Names: RLY-4008

SUMMARY:
The goal of this clinical trial is to evaluate if lirafugratinib is efficacious and safe to treat adult patients with previously treated, unresectable, locally advanced or metastatic solid tumors (excluding cholangiocarcinoma) harboring FGFR2 fusion or rearrangement.

Participants will:

* Take lirafugratinib regularly as instructed by their study doctor.
* Visit the clinic as instructed for checkups and tests.
* Keep a diary recording each time a dose of lirafugratinib is taken.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, locally advanced, or metastatic solid tumor (other than CCA).
* Documented FGFR2 gene fusion or rearrangement per local testing of blood and/or tumor.
* Patient must have measurable disease per RECIST v1.1• Patient has ECOG performance status of 0-1.
* Previously (>30 days) treated with ≥1 line of systemic therapy including chemotherapy (e.g., gemcitabine/cisplatin), immunotherapy, radiation therapy, or other approved therapies.
* Subject has not received prior treatment with an FGFRi.

Exclusion Criteria:

* An uncontrolled comorbidity.
* Patient does not have adequate organ function (defined in protocol).
* Patient has active infection, including human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV) (defined in protocol). Patients with well-controlled HBV are eligible (defined in protocol).
* QT interval corrected using Fridericia's formula (QTcF) > 480 msec or history of prolonged QT syndrome, Torsades de pointes or familial history of prolonged QT syndrome.
* Clinically significant, uncontrolled cardiovascular disease.
* CNS metastases or primary CNS tumor that is associated with progressive neurologic symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by Independent Review Committee per RECIST v1.1. | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months.

SECONDARY OUTCOMES:
Duration of response (DOR) assessed by Independent Review Committee per RECIST v1.1. | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months.
Number of patients with adverse events and serious adverse events. | Every cycle (4-week cycles) until study discontinuation, approximately 24 months.
Number of patients with dose interruptions. | Every 28-day cycle until end of treatment, approximately 24 months.
Number of patients with dose reductions. | Every 28-day cycle until end of treatment, approximately 24 months.
Number of patients with dose discontinuations. | Every 28-day cycle until end of treatment, approximately 24 months.
Objective Response Rate (ORR) as assessed by Investigator per RECIST v1.1. | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months.
Duration of Response (DOR) as assessed by Investigator per RECIST v1.1. | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Disease control rate (DCR) as assessed by Investigator and Independent Review Committee per RECIST v1.1. | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months.
Progression-free survival (PFS) as assessed by Investigator and Independent Review Committee per RECIST v1.1. | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Overall survival (OS). | Up to approximately 36 months.
Time to response (TTR) assessed by Investigator and Independent Review Committee per RECIST v1.1. | Up to approximately 36 months.
Time to progression (TTP) assessed by Investigator and Independent Review Committee per RECIST v1.1. | Up to approximately 36 months
Pharmacokinetic parameters including maximum plasma drug concentration (Cmax) | [Time Frame: Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through Cycle 4 (4-week cycles)]
Pharmacokinetic parameters including area under the plasma concentration versus time curve (AUC) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through Cycle 4 (4-week cycles)
Pharmacokinetic parameters including half-life (t1/2) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through Cycle 4 (4-week cycles)
Change from baseline in quality of life as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). | Approximately every 4 weeks during treatment, approximately 24 months
  It scores (0-100) where higher means better function/quality of life in that section of the questionnaire and higher means worse symptoms in that section of the questionnaire.
Time to deterioration (TTD). | Up to approximately 36 months.
FGFR2 gene status in plasma circulating tumor deoxyribonucleic acid (ctDNA) and tumor tissue. | Every cycle (4-week cycles) through Cycle 3 and every other cycle thereafter until study discontinuation, approximately 24 months.
Pharmacodynamic parameters including changes in fibroblast growth factor 23 (FGF-23). | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every other cycle (4-week cycles) from Cycle 3, approximately 24 months.
Pharmacodynamic parameters including changes in carcinoembryonic antigen (CEA) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every other cycle (4-week cycles) from Cycle 3, approximately 24 months
Pharmacodynamic parameters including changes in cancer antigen 19-9 (CA 19-9) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every other cycle (4-week cycles) from Cycle 3, approximately 24 months
Correlation between FGFR2 genotype by central tissue assessment and antitumor response, as measured by Objective Response Rate (ORR). | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (8):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Gustave Roussy Cancer Campus, Paris
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - START Barcelona-Hospital HM Nou Delfos, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz- START MADRID, Madrid
  - Hospital Universitario HM Sanchinarro-START MADRID-CIOCC, Madrid
- Sarah Cannon Research Institute UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No